CLINICAL TRIAL: NCT02214641
Title: Diabetes Self-Management Lifestyle Intervention for Urban Minority Young Adults
Brief Title: Resilient, Empowered, Active Living: REAL Diabetes Study
Acronym: REAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Beth Pyatak, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1K01DK099202-01A1 (NIH); 1K01DK099202-01A1 (NIH)
Record Dates: First submitted 2014-08-08; First posted 2014-08-12 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle intervention (Experimental): Resilient, Empowered, Active Living (REAL) Diabetes
  Interventions: Behavioral: Resilient, Empowered, Active Living with Diabetes
- Information Control (Active Comparator): Participants will receive a packet of informational materials about diabetes, and receive periodic follow-up phone calls to match for attention dose.
  Interventions: Behavioral: Information Control

INTERVENTIONS:
Behavioral: Resilient, Empowered, Active Living with Diabetes — Individualized lifestyle intervention incorporating the following topics: Diabetes knowledge; access to healthcare; communication with healthcare providers; incorporation of diabetes self-care tasks within daily habits and routines; social support; and emotional well-being. Participants receive a total of 10-16 hours of intervention by a licensed occupational therapist with training in diabetes education, motivational interviewing and the REAL Diabetes intervention protocol.
  Arms: Lifestyle intervention
Behavioral: Information Control — Participants will receive a packet of informational materials about diabetes, and receive periodic follow-up phone calls to match for attention dose. The packet of materials will be delivered in an initial home visit. Follow-up phone calls will occur at approximately two week intervals to inquire whether participants have reviewed specific sections of the intervention materials, and clarify information included in the packet.
  Arms: Information Control

SUMMARY:
This three-year award will pilot-test an innovative intervention, Resilient, Empowered, Active Living with Diabetes (REAL), targeting underserved minority young adults with poorly-controlled diabetes. The individually tailored, community-based intervention merges findings of an in-depth needs assessment, principles of an evidence-based occupational therapy intervention (Lifestyle Redesign®) and evidence-based diabetes self-management strategies. A proof-of-concept study demonstrated that REAL is feasible to implement, acceptable to young adults with type 1 diabetes and type 2 diabetes, and has potential to produce positive changes in diabetes self-care and glycemic control. The study will randomize 80 young adults with diabetes to receive either the six-month REAL intervention or an attention control condition. Blinded data collectors will assess glycemic control, diabetes self-care behaviors and quality of life outcomes, as well as potential intervention mediators, before and after the six-month intervention. It is anticipated that findings from this pilot study will be used to inform a large-scale randomized controlled trial of the REAL intervention.

The study's specific aims and hypotheses are as follows:

Aim 1. Determine the intervention's efficacy for the primary outcomes: glycemic control and diabetes self-care.

Hypothesis: At 6 months (immediately following the intervention), intervention group participants will demonstrate improvements in A1C and diabetes self-care as compared to control group participants.

Aim 2. Conduct exploratory analyses of the intervention's impact on secondary outcomes and potential mediating mechanisms (to inform power estimates for a large-scale RCT).

Hypothesis 1: At 6 months, intervention group participants will demonstrate improvements in secondary outcomes: diabetes-related stress and quality of life, depression, and life satisfaction as compared to control group participants.

Hypothesis 2: At 6 months, intervention group participants will demonstrate improvements in potential mediators of the intervention: habit strength, problem solving, activity participation, self-efficacy and diabetes knowledge as compared to baseline.

Aim 3. Conduct a process evaluation utilizing mixed methods to evaluate and refine intervention delivery (e.g. treatment fidelity, patient satisfaction) and study procedures (e.g. recruitment, retention, testing protocol).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 or type 2 diabetes mellitus for a minimum of 12 months
* Most recent A1C ≥8.0%
* Fluent in English or Spanish
* Reachable by telephone or text message
* Willing to participate in study activities
* Reside in Los Angeles County with no plans to relocate

Exclusion Criteria:

* Pregnant or planning to become pregnant
* Cognitive impairment or severe disability limiting life expectancy
* Participated in lifestyle intervention targeting diabetes within past 12 months
* Participated in formative research related to intervention development.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1C) | Baseline & 6 months.
  Measure of average blood glucose concentration over approximately the previous 12 weeks.

SECONDARY OUTCOMES:
Audit of Diabetes-Dependent Quality of Life (ADD-QoL) | Baseline & 6 months.
  19-item survey measure assessing impact of diabetes on social, physical, and emotional functioning.
Problem Areas in Diabetes (PAID) Scale - Short Form | Baseline & 6 months.
  5-item survey measure assessing diabetes-related distress and emotional problems.
Patient Health Questionnaire-8 (PHQ-8) | Baseline & 6 months
  8-item survey measure assessing severity of depressive symptoms (identical to PHQ-9 while omitting self-harm item).
Satisfaction With Life Scale (SWLS) | Baseline & 6 months.
  5-item survey measure assessing global life satisfaction and subjective well-being.
Summary of Diabetes Self-Care Activities (SDSCA) | Baseline & 6 months
  14 items assessing diet, physical activity, medication adherence and other self-care behaviors relevant to diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Pyatak, PhD, OTR/L, Principal Investigator — University of Southern California
Locations (1):
- USC, Los Angeles, California, United States

REFERENCES:
- [Background] Pyatak EA, Florindez D, Peters AL, Weigensberg MJ. "We are all gonna get diabetic these days": the impact of a living legacy of type 2 diabetes on Hispanic young adults' diabetes care. Diabetes Educ. 2014 Sep-Oct;40(5):648-58. doi: 10.1177/0145721714535994. Epub 2014 May 27. PMID 24867918
- [Background] Pyatak EA, Sequeira PA, Whittemore R, Vigen CP, Peters AL, Weigensberg MJ. Challenges contributing to disrupted transition from paediatric to adult diabetes care in young adults with type 1 diabetes. Diabet Med. 2014 Dec;31(12):1615-24. doi: 10.1111/dme.12485. Epub 2014 May 26. PMID 24798586
- [Background] Pyatak EA, Florindez D, Weigensberg MJ. Adherence decision making in the everyday lives of emerging adults with type 1 diabetes. Patient Prefer Adherence. 2013 Jul 29;7:709-18. doi: 10.2147/PPA.S47577. Print 2013. PMID 23935361
- [Background] Pyatak EA, Carandang K, Davis S. Developing a Manualized Occupational Therapy Diabetes Management Intervention: Resilient, Empowered, Active Living With Diabetes. OTJR (Thorofare N J). 2015 Jul;35(3):187-94. doi: 10.1177/1539449215584310. PMID 26594741
- [Background] Pyatak EA, Carandang K, Vigen C, Blanchard J, Sequeira PA, Wood JR, Spruijt-Metz D, Whittemore R, Peters AL. Resilient, Empowered, Active Living with Diabetes (REAL Diabetes) study: Methodology and baseline characteristics of a randomized controlled trial evaluating an occupation-based diabetes management intervention for young adults. Contemp Clin Trials. 2017 Mar;54:8-17. doi: 10.1016/j.cct.2016.12.025. Epub 2017 Jan 5. PMID 28064028
- [Background] Vigen CLP, Carandang K, Blanchard J, Sequeira PA, Wood JR, Spruijt-Metz D, Whittemore R, Peters AL, Pyatak EA. Psychosocial and Behavioral Correlates of A1C and Quality of Life Among Young Adults With Diabetes. Diabetes Educ. 2018 Dec;44(6):489-500. doi: 10.1177/0145721718804170. Epub 2018 Oct 8. PMID 30295170
- [Background] Carandang KM, Pyatak EA. Feasibility of a Manualized Occupation-Based Diabetes Management Intervention. Am J Occup Ther. 2018 Mar/Apr;72(2):7202345040p1-7202345040p6. doi: 10.5014/ajot.2018.021790. PMID 29426394
- [Result] Pyatak EA, Carandang K, Vigen CLP, Blanchard J, Diaz J, Concha-Chavez A, Sequeira PA, Wood JR, Whittemore R, Spruijt-Metz D, Peters AL. Occupational Therapy Intervention Improves Glycemic Control and Quality of Life Among Young Adults With Diabetes: the Resilient, Empowered, Active Living with Diabetes (REAL Diabetes) Randomized Controlled Trial. Diabetes Care. 2018 Apr;41(4):696-704. doi: 10.2337/dc17-1634. Epub 2018 Jan 19. PMID 29351961
- [Derived] Salvy SJ, Carandang K, Vigen CL, Concha-Chavez A, Sequeira PA, Blanchard J, Diaz J, Raymond J, Pyatak EA. Effectiveness of social media (Facebook), targeted mailing, and in-person solicitation for the recruitment of young adult in a diabetes self-management clinical trial. Clin Trials. 2020 Dec;17(6):664-674. doi: 10.1177/1740774520933362. Epub 2020 Jul 6. PMID 32627589